CLINICAL TRIAL: NCT07132502
Title: Treatment Intermittent Periods Based on ctDNA-MRD Status in Advanced HER2-Positive Breast Cancer: A Non-Interventional Exploratory Study
Brief Title: Treatment Intermittent Periods Based on ctDNA-MRD（Circulating Tumor DNA-minimal Residual Disease） Status in Advanced HER2-Positive Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, PENG YUAN, Department Director, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NC5269
Record Dates: First submitted 2025-07-06; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: ctDNA MRD — Definition and Essence: ctDNA MRD involves detecting DNA fragments released by tumor cells into the bloodstream through highly sensitive techniques to determine the status of minimal residual disease in cancer patients.
  Detection Methods: Technologies such as digital PCR and next-generation sequencing (NGS) are employed to achieve precise detection of low-frequency ctDNA mutations.
  Clinical Significance: It is utilized for evaluating the prognosis of cancer patients and providing crucial evidence for the formulation of personalized treatment plans.

SUMMARY:
Breast cancer seriously threatens the health of women worldwide. The HER-2-positive subtype accounts for approximately 15% to 20%, featuring strong invasiveness and poor prognosis. In recent years, anti-HER-2 targeted therapy has developed rapidly. The application of various drugs has improved the remission rate of advanced patients, leading to an increase in the number of patients achieving complete remission (CR). However, CR patients still face the risk of recurrence. Moreover, treatment decisions are confronted with dilemmas such as the contradiction between the cumulative toxicity of continuous treatment and the increased risk of recurrence due to premature drug withdrawal, as well as the lack of step-down treatment guidance strategies in disease-free states.

Circulating tumor DNA (ctDNA)-mediated molecular residual disease (MRD) detection shows potential in predicting prognosis and monitoring recurrence in various solid tumors, with certain progress also made in the field of breast cancer. However, there are few studies on its application in guiding treatment decisions for advanced HER-2-positive breast cancer patients after CR.

This study adopts a prospective, observational cohort study design. It intends to screen advanced HER-2-positive breast cancer patients, include those who have achieved CR with negative ctDNA-MRD and negative CA153, and divide them into a drug intermission group and a continued salvage treatment group based on patients' autonomous choices. The study will conduct long-term follow-up on the two groups, dynamically monitor the ctDNA-MRD status, observe the disease changes when treatment is paused in the drug intermission group, as well as the treatment response and disease progression in the continued salvage treatment group. It will evaluate the impact of the drug intermission strategy on prognostic indicators such as progression-free survival (PFS) and overall survival (OS), clarify whether ctDNA-MRD can accurately predict recurrence risk to guide individualized treatment, explore the feasibility and safety of the drug intermission strategy to balance efficacy and toxicity, screen patients with good prognosis to provide a basis for step-down treatment, and promote precision treatment for advanced HER-2-positive breast cancer, filling the research gap.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed HER-2 positive breast cancer (immunohistochemistry 3+ or 2+ with FISH positivity).Diagnosis of advanced breast cancer in accordance with AJCC staging criteria.
* Achieved complete response (CR) as evaluated by PET-CT or contrast-enhanced CT after receiving salvage therapy (within second-line) and maintained for 3 months.
* Negative ctDNA-MRD (circulating tumor DNA - minimal residual disease) detection.
* Negative CA153 detection.
* ECOG performance status score of 0-2.
* Expected survival ≥ 6 months.
* The patient has signed an informed consent form, willing to cooperate with the study and accept regular follow-up.

Exclusion Criteria:

* Concomitant other malignant tumors (excluding breast cancer).
* History of mental disorders or cognitive dysfunction, unable to cooperate with the study.
* Pregnant or lactating women.
* Severe cardiac, hepatic, or renal insufficiency.
* Currently participating in other clinical trials that may affect the evaluation of this study's results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population refers to patients with advanced HER-2 positive breast cancer who have achieved complete response (CR), negative ctDNA-MRD (circulating tumor DNA - minimal residual disease), and negative CA153.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2027-07-08 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Progression - free survival (PFS) | from July 2025 to June 2027

SECONDARY OUTCOMES:
Overall survival (OS): | from July 2025 to June 2027
Treatment - free interval | from July 2025 to June 2027
Patient quality of life assessment | from July 2025 to June 2027
  specific quality of life scales such as EORTC QLQ - C30 （European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30）1.Functional domains (e.g., physical functioning, emotional functioning, etc.): A higher score indicates better functioning in that aspect (e.g., a score of 100 represents fully normal functioning, while a score of 0 indicates severe functional impairment).
  2.Symptom domains (e.g., fatigue, pain, etc.) and global quality of life domain: For symptom domains, a higher score indicates more severe symptoms or poorer quality of life; for the global quality of life domain, a higher score indicates better overall quality of life.

IPD SHARING:
Plan to Share IPD: Undecided